CLINICAL TRIAL: NCT03999671
Title: Effect of the Nursing Process Through Functional Patterns on the Quality of Life of the Elderly Adult Patient With Definitive Pacemaker Implantation
Brief Title: Effect of the Nursing Process on the Quality of Life of the Patient With Definitive Pacemaker Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Sonia Gonzalez Mejorada, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R-2013-3604-7
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Quality of Life
Keywords: Effect, Nursing, Process, Functional, Patterns,health

STUDY DESIGN:
Intervention Model Description: Control group and intervention group, were selected randomly from consecutive cases and standard management
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INSTRUMENT SF 36 (Experimental): Instrument SF36 Spanish version, validated in Spain, translated in several languages and applied to multiple studios in Mexico. The 36 items explore 8 dimensions: the state of physical health, physical function, physical role, body pain, general health, vitality, social function, emotional role and mental health: considering depression, anxiety, self-control, and general well-being.
  Interventions: Other: Educational; Other: Maneuver control
- Checklist (Active Comparator): Verify that the interventions of both groups were carried out
  Interventions: Other: Educational; Other: Maneuver control

INTERVENTIONS:
Other: Educational — Traditional method of nursing care with what is done every day, with the method through the nursing process using nursing language as a nursing diagnosis, classification of nursing interventions, and nursing outcomes.
Other: Maneuver control — Verify that the control and intervention group developed the assigned activities in each case.

SUMMARY:
The nursing process consists of establishing interventions applying the scientific method for the resolution of real or potential health problems of the person, based on five stages: assessment, diagnosis, planning, execution and evaluation, which allows detecting the circumstances and elements that affect the adult's independence and the influence he has on his environment, his quality of life, his family, social and psychological role.

MATERIAL AND METHODS: Clinical trial, randomized, controlled with standard management; to evaluate the effect of the nursing process on the quality of life in elderly patients who come or are referred to the Cardiology Hospital, National Medical Century XXI, with alterations in the ventricular atrial conduction and require the installation of a permanent pacemaker. The first evaluation (Time 0) will be carried out through an interview with the SF36 instrument, translated into several languages and applied to multiple studies in Mexico for validation. Two groups will be formed for comparison: Group I will be assigned to standard management; Group II: group of patients who are also treated through the nursing process with the model of Marjory Gordon with the intervention Handling the definitive pacemaker with education and information activities. It will be verified for quality control of the maneuver; through a checklist. As a final point, the quality of life will be evaluated through the use of the SF36 instrument that consists of 36 items that explore 8 dimensions of the state of physical health, physical function, physical role, body pain, general health, vitality, social function, emotional role and mental health: considering depression, anxiety, self-control, and general well-being; applying the assessment system of the functional patterns of the Marjory Gordon model, through surveys. Statistical analysis: Chi square or Fisher's exact test will be used according to expected values, for qualitative variables. For quantitative variables, the Mann Whitney U or Student's T according to their distribution. There will be a calculation of the number needed to be treated, and a multivariate analysis will be carried out using a binary logistic regression.

DETAILED DESCRIPTION:
Patients admitted to the Cardiology Hospital, National Medical Center Century XXI, will be included and a permanent pacemaker will be installed due to alterations in atrio-ventricular conduction that meet the selection criteria. They will be explained what the research consists of and they will be given an informed consent form to participate in the study, with all the ethical considerations that we will discuss later.

they require to control their comorbidities according to the assessment of their treating physician. Having accepted their participation in the present research project, the first evaluation (Time 0) will be conducted through an interview with the instrument SF36 Spanish version containing a total of 36 questions, translated into several languages and applied to multiple studies in Mexico for its validation. The interview will be conducted in two parts and will last approximately 15 to 20 minutes.

Once the first evaluation has been carried out, they will randomly assign, through the use of random number tables, to receive specific care from the nursing staff in the following manner:

I. Group of conventional nursing intervention (Group I) that refers to the form performed up to now, hemodynamic assessment, local pacemaker verification, electrocardiographic tracing, surveillance and care of the incision, assessment of symptoms after the insertion of the pacemaker, risks and interferences, mobilization and posture, complications, care information and identification of other needs of the elderly in terms of mobility, degree of dependency, pain assessment, elimination, nutritional, rest and relationship difficulties family, work, emotional conflicts, values and religiosity in some cases.

II. Nursing intervention group through the nursing process with the Marjory Gordon system (Group II).

1. Starting with the assessment stage by functional patterns: health perception-management, nutrition, elimination, activity and rest, sleep and rest, perceptual cognitive, self-concept-self-perception, role-relationships, sexuality-reproduction, coping-tolerance of stress, values and beliefs and the quality of life.
2. Following the diagnostic stage of nursing, the problem is identified through labels that define it as: Decrease in cardiac output, risk of bleeding, ineffective protection, acute pain, risk of imbalance of body temperature, deterioration of ambulation, deterioration of physical mobility, deterioration of gas exchange, disposition to improve one's health, sleep deprivation, deterioration of urinary elimination, constipation, self-care deficit, sensory perception disorder, deterioration of social interaction or conflict of decisions , hopelessness, low self-esteem, body image disorder, ineffective coping, anxiety, fear and hopelessness complementing the structure of the diagnosis with risk factors (for example: poor knowledge) and etiological (for example: altered frequency and heart rate) , as well as, with defining characteristics (signs and symptoms) that pre Say the problem.
3. The planning stage will be carried out through expected results from the problems identified as nursing diagnoses and using the classification of expected nursing outcomes (NOC) each of them with a target score of maintaining results; will increase; and scales from severe to none, or from seriously compromised to uncommitted will depend on the proposed result. Decreased cardiac output The expected result will be effectiveness of the heart pump which will be measured with indicators such as: systolic blood pressure, diastolic blood pressure, heart rate , peripheral pulses. From the expected result, nursing interventions will be derived:

   Intervention "Cardiac care" with activities
   1. Observing vital signs frequently
   2. Monitor cardiovascular status
   3. Check and check the operation of the pacemaker,
   4. Instruct the patient on the importance of the immediate report of any chest discomfort.
   5. Take note of the significant signs and symptoms of decreased cardiac output. • Intervention "Management of the definitive pacemaker" with activities of

   <!-- -->

   1. Education on the potential risks of metabolic alterations (eg potential to increase the thresholds of rhythm or capture);
   2. The importance of attending their periodic checks;
   3. Sources of higher electromagnetic interference (eg arc welding equipment, radio transmitters, electronic muscle stimulators, concert loudspeakers, electric drills, hand-held metal detectors, magnetic resonance, radiotherapy).
   4. Keep about 15 cm away from cell phones;
   5. Signs and symptoms of a dysfunctional pacemaker (eg bradycardia, dizziness, weakness, fatigue, chest discomfort, angina, dyspnea, orthopnea, edema, paroxysmal nocturnal dyspnea, exertional dyspnea, hypotension, syncope, cardiac arrest)
   6. The importance of carrying the identification card of the manufacturer at all times.
   7. Information to the patient and the family related to the implantation of the pacemaker (eg, indications, functions, universal programming codes, potential complications); related to the effects of pacemaker treatment to reduce patient uncertainty, fear and anxiety about symptoms (eg dizziness, palpitations, chest pain, shortness of breath) related to treatment (arm edema or augmentation) of heat);
   8. Teach the patient to check the manufacturer's warnings when in doubt about electrical appliances.
4. Fourth stage of the nursing process execution of nursing interventions (NIC) obtained through the expected results (NOC).

To evaluate the response of patients to nursing interventions in their quality of life, the following will be done:

1. Before discharge from hospital, verification of quality control of the maneuver will be carried out, using a checklist, on the indications given by the nursing staff to the patient.

2. One month after the patient's hospital discharge, during which patients are regularly scheduled for follow-up consultation, after their routine medical assessment, an interview will be conducted where we will make a total of 36 questions with 3 to 5 answer options each, with the SF36 instrument. The 36 items explore 8 dimensions of the state of physical health, physical function, physical role, body pain, general health, vitality, social function, emotional role and mental health: considering depression, anxiety, self-control, and general well-being; applying the assessment system of the functional patterns of the Marjory Gordon model, through surveys. The interview will be conducted in two parts and will last approximately 15 to 20 minutes. (Outcome) The system by Functional Employers focuses its attention on 11 items with importance for the health of the individual, family or community.

1. Ability of the person to identify their health status.
2. Ability of the person to identify their nutritional needs.
3. Identify the excretory function (intestinal, urinary and skin).
4. Realization of the activities and exercise carried out by the person.
5. Conciliar sleep activity
6. Sensory alterations: Hearing, gustatory, tactile and olfactory views as well as the presence of pain.
7. Form in which the patient feels, feelings, knowledge of himself.
8. Way to live with others.
9. It is experienced or expressed in the form of thoughts, fantasies, desires, beliefs, attitudes, values, activities, practices, roles and relationships.
10. Way to handle stress.
11. Values, beliefs that guide the decisions and choices of the individual.

ELIGIBILITY:
Inclusion criteria:

* Adults over 60 years old
* Any gender
* That require the placement of a definitive pacemaker either by endocardial or epicardial route and do not present any complication during its installation and hospital stay.
* Signature of informed consent in writing of acceptance to enter the study

Exclusion criteria:

* Older adults with neurological problems.
* Patients with other aggregate pathologies different from atrio-ventricular conduction abnormalities such as valvular diseases, myocardial infarction, congenital diseases, postoperative atrio-ventricular blocks, neoplastic diseases, end-stage renal disease.
* Generator depletion.
* Endocarditis.
* Chronic degenerative diseases whose life expectancy is less than 2 years.
* Previous pacemaker carrier and that you enter for replacement.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Effect of the Nursing Process Through Functional Patterns on the Quality of Life of the Elderly Adult Patient With Definitive Pacemaker Implantation | one year
  To determine the effect of the nursing process through the functional patterns on the quality of life of the elderly adult patient with definitive pacemaker implantation.

CONTACTS AND LOCATIONS:
Overall Officials: SONIA GONZALEZ MEJORADA, Principal Investigator — Instituto Mexicano del Seguro Social